CLINICAL TRIAL: NCT01347450
Title: Protective Effects of Cocoa Ingestion Over Healthy Males Plasma Lipids Subjected to Peroxidative Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Santa Fe de Bogota (Other)
Collaborators: Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government)
Responsible Party: Manuel Barrios, Fundación Santa Fe de Bogotá
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 20114
Record Dates: First submitted 2011-04-29; First posted 2011-05-04 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2004-09

CONDITIONS: Lipid Peroxidation
Keywords: Flavonoids; cacao; lipid peroxidation; plasma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cocoa, Placebo (Experimental)
  Interventions: Dietary Supplement: Cocoa powder berverage, dark chocolate bar; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cocoa powder berverage, dark chocolate bar — Sugar drink containing 30 g of cocoa powder and 50 g of a 65% dark chocolate, and the control group received 30 g of placebo drink containing 0 g of cocoa powder. Each drink was prepared by using 300 ml of water and 30 g of sugar, also were consumed twice each day: with breakfast and afternoon meal. during 7-d after the intervention started.
Dietary Supplement: Placebo — Sugar drink containing 30 g of cocoa powder and 50 g of a 65% dark chocolate, and the control group received 30 g of placebo drink containing 0 g of cocoa powder. Each drink was prepared by using 300 ml of water and 30 g of sugar, also were consumed twice each day: with breakfast and afternoon meal. during 7-d after the intervention started.

SUMMARY:
Background: Cocoa is rich in flavonoids such as (-)-epicatechin and (+)-catechin; these compounds have displayed both in vitro and in vivo antioxidant activity.

Objective: This trial evaluate the regular ingestion effect of both, dark chocolate and cocoa powder, over plasma lipids of young males subjected to ex vivo lipid peroxidative conditions.

Design: Single-blind, controlled and randomized clinical trial including 100 healthy men, divided into two groups: 50 subjects received 30 g of cocoa powder and 50 g of dark chocolate/d for 1 wk, and the other 50 subjects received placebo.

DETAILED DESCRIPTION:
Adult young males were enrolled at the Universidad Industrial de Santander by publicity at the university food service centre. Those who respond (n=136) were selected after the normal blood lipid profile was verified by laboratory testing of total cholesterol, LDL, HDL, VLDL and triacylglycerols, as well exclusion and inclusion criteria were applied. Within the exclusion criteria we included diagnosed coronary artery disease, diabetes mellitus, arterial hypertension, use of any prescribed medication, restrictive diets and any migraine or cocoa products allergic antecedents.

Finally enlisted subjects were 120 non-smokers, normolipemic, ages were between 20 and 30 years old, who underwent anthropometric measurements like weight, height, BMI (among 16.0 and 27.4 kg/m2) and regular nutritional and toxicological habits using standardized surveys. Subjects received 3 meals a day from the Food Nutritional Service of Universidad Industrial de Santander, in order to ensure the same diet conditions for all subjects along the experimental period. An average colombian diet, based on 2287 calories as a total caloric value (protein 15%, fats 35% and carbohydrates 60%) was used. The study protocol and the informed consent were approved by the Fundación Santa Fe de Bogotá Institutional Ethical Committee (Santa Fe de Bogotá D.C., Colombia). We got written informed consent from all participants and they received money compensation for its participation in the study.

Outcome measures:

Susceptibility of plasma lipids to oxidation Determination of plasma lipids oxidation resistance Determination of oxidative protection

ELIGIBILITY:
Inclusion Criteria:

* Normal lipid profile
* Age between 20 and 30 years old
* Must like chocolate

Exclusion Criteria:

* Diagnosed coronary artery disease
* Diabetes mellitus
* Hypertension
* Use of any prescribed medication
* Restrictive diets and any
* Migraine or
* Cocoa products allergic antecedents

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2007-10; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Oxidative protection index | 7-days after the intervention started.
  Oxidative protection of plasma lipids was set up by measuring hexanal, known as one of the main components of oxidizing n-6 polyunsaturated fatty acids (PUFA). The oxidative protection index (OPI), was defined as the difference between the basal and post intervention (cocoa taking in) sample chromatographic areas as stated by the formula: OPI = (Area0 - Area1/ Area0)*100. Hexanal determination was carried out by HS-SPME in situ derivatization method using PFPH fibre saturation as derivatizing agent under the methodology

SECONDARY OUTCOMES:
Oxidation resistance index (ORI) | 7-days after the intervention started
  ORI was expressed as a percentage and held as the difference among basal (0) and post interventions (1) lag time of each subject according to the following formula: ORI = (lag1 - lag0/ lag1)*100. Plasma was 50-fold diluted in a saline phosphate solution (PBS; 0.0027M KCl, 0.137M NaCl, pH 7.4) and then was exposed to copper (II) chloride at final concentration of 95 µM in a 2.5 ml quartz cuvette. Conjugated diene formation from lipid peroxidation was followed at 245 nm wavelength, recorded each 5 min over 4-h period at 37ºC in a Perkin Elmer Lambda Bio 10 spectrophotometer

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Carrasquilla, PhD, Study Director — Fundación Santa Fe de Bogotá
Locations (1):
- Fundación Santa Fe de Bogotá, Universidad Industrial de Santander., Bogotá DC., Bogotá DC., Colombia

REFERENCES:
- [Derived] Barrios M, Orozco LC, Stashenko EE. Cocoa ingestion protects plasma lipids in healthy males against ex vivo oxidative conditions: A randomized clinical trial. Clin Nutr ESPEN. 2018 Aug;26:1-7. doi: 10.1016/j.clnesp.2018.05.001. Epub 2018 May 30. PMID 29908675